CLINICAL TRIAL: NCT00514085
Title: A Phase II Study of Interleukin-21 (IL-21) in Patients With Metastatic or Recurrent Malignant Melanoma
Brief Title: Interleukin-21 in Treating Patients With Metastatic or Recurrent Malignant Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: ZymoGenetics (Industry)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I189; CAN-NCIC-IND189 (Registry Identifier: NCI US - Physician Data Query); IND.189 (Other: NCIC CTG Trial Identifier); ZYMOGENETICS-CAN-NCIC-IND189 (Other: Zymogenetics); CDR0000560973 (Other: PDQ)
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Recombinant human interleukin-21 (Experimental)
  Interventions: Biological: recombinant human interleukin-21; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Biological: recombinant human interleukin-21 — Patients enrolled in Part A will receive treatment daily x 5 on weeks 1, 3, and 5 of an 8 week cycle.
  Patients enrolled in Part B will receive treatment daily x 5 on weeks 1, and 3 of a 6 week cycle
Other: immunohistochemistry staining method — Cycle 1 Day 1 and Cycle 1 Day 29
Other: laboratory biomarker analysis — slides will be blocked for 15 minutes in 20% normal goat serum and then incubated in primary antibody
Other: pharmacological study — Starting dose of 50μg/kg/day as an IV push

SUMMARY:
RATIONALE: Interleukin-21 may stimulate white blood cells, including natural killer cells, to kill melanoma cells.

PURPOSE: This phase II trial is studying the side effects and how well interleukin-21 works in treating patients with metastatic or recurrent malignant melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the efficacy, in terms of objective response rate, nonprogression rate, time to progression, and response duration, in patients with metastatic or recurrent malignant melanoma treated with recombinant human interleukin-21 (rIL-21).
* To assess the toxicity and safety of rIL-21 in patients with previously untreated metastatic or recurrent malignant melanoma.
* To characterize the pharmacokinetics of rIL-21.
* To characterize the effects of rIL-21 on lymphocyte cell count and soluble CD25 (sCD25) in serum as potential biomarkers for drug activity.
* To evaluate the immunogenicity of rIL-21, specifically preexisting immunogenicity to the drug and antibody induction during treatment.
* To assess melanoma antigenic markers for response and nonprogression on archival tissue from patients enrolled on the study.

Secondary

* To investigate whether rIL-21 induced sCD25 release is independent of the level of circulating sCD25.
* To investigate the effect of rIL-21 on antibody induction during treatment and preexisting immunogenicity.
* To assess lymphocyte cell-count changes over time in relation to rIL-21 therapy.

OUTLINE: This is a multicenter study.

Patients receive recombinant human interleukin-21 (rIL-21) IV on days 1-5 of weeks 1, 3 and 5. Treatment repeats every 8 weeks in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) or partial response (PR) receive 2 courses beyond CR or PR. Patients with stable disease receive a maximum of 3 courses of rIL-21.

Previously archived tumor tissue and blood samples are collected from patients for correlative studies. Samples are analyzed for soluble CD25, rIL-21 antibodies, circulating lymphocyte counts, preexisting immonogenicity to rIL-21 for antibody induction, and expression of common melanoma tumor antigen markers via IHC.

After completion of study treatment, patients are followed at 4 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cutaneous malignant melanoma

  * Recurrent or metastatic disease that is not curable by surgical or other means
* Clinically and/or radiologically documented disease defined as at least one site of disease unidimensionally measurable ≥ 20 mm by x-ray, physical exam, or nonspiral CT scan OR ≥ 10 mm by spiral CT scan
* Must have nonbulky metastatic disease defined as the largest measurable lesion ≤ 50 mm in maximum diameter
* Must have primary diagnosis tumor tissue or previously resected metastatic melanoma tissue available (i.e., paraffin block or unstained slides)
* No known brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* Absolute granulocytes count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin normal
* Serum creatinine ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Negative pregnancy test
* Not pregnant or nursing
* Fertile patients must use effective contraception during study therapy
* No uncontrolled intercurrent illness or condition including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situation that would limit compliance with study requirements
* No history of hemolysis or a hemolytic disorder including, but not limited to, any of the following:

  * Sickle cell anemia
  * Thalassemia
  * Autoimmune hemolytic anemia
* No history of other malignancies within the past 5 years except adequately treated nonmelanoma skin cancer, curatively treated carcinoma in situ of the cervix, or other solid tumors curatively treated with no evidence of disease
* No known HIV, hepatitis B, or hepatitis C infection
* Patients must reside within a 2-hour drive from a participating center

PRIOR CONCURRENT THERAPY:

* No previous systemic therapy for metastatic disease
* At least 3 months since prior adjuvant immunotherapy for recurrent melanoma

  * No prior immunotherapy for metastatic disease
  * No prior immunotherapy outside the adjuvant setting
* At least 4 weeks since prior major surgery
* At least 4 weeks since prior radiotherapy except low-dose, nonmyelosuppressive radiotherapy and recovered
* More than 4 weeks since prior and no concurrent investigational agents or anticancer therapy
* No prior chemotherapy including regional therapy
* No concurrent systemic corticosteroids (e.g., prednisone or dexamethasone)

  * Concurrent topical steroids are allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-12-13 (Actual); Primary Completion 2010-09-02 (Actual); Study Completion 2012-07-04 (Actual)

PRIMARY OUTCOMES:
Objective tumor response as assessed by RECIST | after completion of treatment
Overall response rate (complete and partial) | after completion of study
Stable disease rate | after completion of study
Progressive disease rate | after completion of study
Median time to progression | after completion of study
Response duration (median and range) | after completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Teresa M. Petrella, Study Chair — Toronto Sunnybrook Regional Cancer Centre
Locations (7):
- Canada (7):
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Petrella TM, Tozer R, Belanger K, Savage KJ, Wong R, Smylie M, Kamel-Reid S, Tron V, Chen BE, Hunder NN, Hagerman L, Walsh W, Eisenhauer EA. Interleukin-21 has activity in patients with metastatic melanoma: a phase II study. J Clin Oncol. 2012 Sep 20;30(27):3396-401. doi: 10.1200/JCO.2011.40.0655. Epub 2012 Aug 20. PMID 22915661